CLINICAL TRIAL: NCT01751230
Title: E-Moms: A Personalized Telehealth Intervention for Health and Weight Loss in Postpartum Women
Brief Title: A Personalized Telehealth Intervention for Health and Weight Loss in Postpartum Women
Acronym: E-Moms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: University of California, Los Angeles (Other); United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Leanne Redman, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PBRC 12030
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Postpartum Weight Retention
Keywords: pregnancy; weight loss
MeSH Terms: conditions — Gestational Weight Gain; Weight Loss

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WIC E-Moms (Experimental): If picked for this group, you will receive a personalized diet and exercise plan to help you lose the weight you gained during your pregnancy. All information will be given to you using a SmartPhone, such as an iPhone. You can use your own phone or one can be loaned to you for the study. You will also be loaned a scale so you can weigh yourself at home. You will also get advice and services from your WIC clinic.
  Interventions: Behavioral: WIC E-Moms
- WIC Moms (No Intervention): You will get advice and services for nutrition and weight management after pregnancy from your WIC clinic.

INTERVENTIONS:
Behavioral: WIC E-Moms — Participants enrolled in the E-Moms group will receive a personalized dietary prescription to promote weight loss and arrive at pregravid weight by 6 months postpartum. Our weight loss intervention will incorporate standard WIC nutritional advice and will encouraged 150 minutes/week of moderate intensity activity, which is about 3,000 - 4,000 steps/day above baseline, as recommended for maintenance of healthy weight. Each participant will be assigned a trained weight management counselor who will provide frequent recommendations and advice and support at least once per week.
  Other Names: E-Moms
  Arms: WIC E-Moms

SUMMARY:
The purpose of this study is to help women lose the weight they gained during their pregnancy using a SmartPhone app the investigators have developed called E-Moms. The investigators hypothesize that the moms given the app to use during the study will lose more weight than the moms who do not use the app.

DETAILED DESCRIPTION:
The E-Moms Study will last about 4 months. The weight management program is 4 months long and will end about 6 months after the participant's baby is born. All participants will receive Women, Infants and Children (WIC) services.

For the weight management program, participants will be put into one of these groups:

1. WIC Moms: receive advice and services for nutrition and weight management after pregnancy from their WIC clinic.
2. WIC E-Moms: receive a personalized diet and exercise plan to help them lose the weight they gained during their pregnancy. All information will be given to them using a SmartPhone, such as an iPhone. They will also get advice and services from your WIC clinic.

ELIGIBILITY:
Inclusion Criteria:

* Are a female who has delivered a baby within the last 2 months
* Are 18 years of age or older
* Have a body mass index ≥25 kg/m2 or <40 kg/m2
* Are accepted for post-pregnancy WIC services
* Are English-speaking

Exclusion Criteria:

* Are participating in the Nurse Family Partnership program
* Had multiples in your most recent pregnancy
* Are unwilling to be assigned at random to either of the 2 study groups
* Are planning to move out of the study area within the next 6 months
* Have a history of psychiatric conditions or chronic disease than can impact body weight, appetite, or energy intake such as HIV/AIDS, cancer, bipolar disorder or schizophrenia
* Currently use antipsychotic medications or have used such medications in the previous 12 months
* Have been diagnosis with type I diabetes
* Report having a heart attack, stroke, or being hospitalized or treated for chest pain
* Currently taking medications or supplements to aid in weight loss
* Have had weight loss surgery in the past year or plan to have it prior to study completion.
* Currently participating in another interventional study that influences weight control
* Currently abusing drugs or alcohol (up to 14 drinks per week allowed)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Redman, M.S., Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
Study data available upon request and following appropriate data transfer agreements in place.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants will be recruited via Institutional Review Board (IRB) approved posters and flyers displayed in the WIC office and advertisements posted on the PBRC website (http://www.pbrc.edu/clinicaltrials).
Groups:
- WIC E-Moms: Participants enrolled in the WIC E-Moms group will receive a personalized dietary prescription to promote weight loss and arrive at pregravid weight by 6 months postpartum. Our weight loss intervention will incorporate standard WIC nutritional advice and will encouraged 150 minutes/week of moderate intensity activity, which is about 3,000 - 4,000 steps/day above baseline, as recommended for maintenance of healthy weight. Each participant will be assigned a trained weight management counselor who will provide frequent recommendations and advice and support at least once per week.
- WIC Moms: Participants in WIC Moms will receive standardized advice and services for postpartum nutrition and weight management through their nominated WIC clinic. Participants in the control group will not receive a dietary prescription or personalized weight management services from the Pennington Biomedical study team.
Period: Overall Study
Arm/Group | WIC E-Moms | WIC Moms
Started | 20 | 20
Completed | 19 | 16
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | WIC E-Moms | WIC Moms | Total
Number analyzed (Participants) | 19 | 16 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.0 (5.2) | 27.2 (6.1) | 26.5 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 35
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 14 | 26
  White | 6 | 2 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Preconception weight [Mean (Standard Deviation); unit: kg] | 80.7 (9.1) | 79.9 (17.4) | 80.4 (14.2)
Gestational weight gain [Mean (Standard Deviation); unit: kg] | 14.3 (9.2) | 15.2 (8) | 14.7 (8.6)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.3 (3.2) | 32.7 (2.8) | 32.1 (3.3)
Enrollment weight [Mean (Standard Deviation); unit: kg] | 83.8 (13.5) | 88.4 (9.7) | 85.9 (12.0)
Body fat [Mean (Standard Deviation); unit: %] | 40.2 (4.7) | 41.7 (3.8) | 40.9 (4.3)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 117.5 (13.8) | 116.7 (12.6) | 117.2 (13.2)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 74.6 (9.2) | 73.9 (10.1) | 74.5 (9.7)
Parity [Mean (Standard Deviation); unit: pregnancies] | 1.6 (1.0) | 2 (1.3) | 1.8 (1.2)
Marital status [Count of Participants; unit: Participants]
  Married | 5 | 3 | 8
  Not married and living with significant other | 6 | 3 | 9
  Separated/divorced | 0 | 1 | 1
  Single | 8 | 9 | 17
Education [Count of Participants; unit: Participants]
  Some high school | 1 | 0 | 1
  High school diploma/General education development | 6 | 3 | 9
  1-3 college | 5 | 9 | 14
  College degree | 5 | 3 | 8
  Postgraduate | 2 | 1 | 3
Breastfeed ever [Count of Participants; unit: Participants]
  No | 4 | 5 | 9
  Yes | 15 | 11 | 26
Current smoker [Count of Participants; unit: Participants]
  No | 18 | 13 | 31
  Yes | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Body Weight Change
Description: The primary outcome measure is weight change after the 16 week intervention.
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Error); unit: kg
Arm/Group | WIC E-Moms | WIC Moms
Number analyzed (Participants) | 19 | 16
kg | -0.1 (0.9) | 1.8 (0.9)

2. Post Hoc Outcome: Changes in Hip Circumference of WIC Moms, WIC E-Moms Subgroups: High, Medium, and Low Adherers
Description: Changes in hip circumference from baseline (Week 0) stratified by adherence to the E-Moms intervention and usual care (WIC Moms).
Time Frame: Baseline and 16 weeks
Population: All participants stratified by adherence to the E-Moms intervention and usual care (WIC Moms)
Measure: Mean (Standard Error); unit: cm
Groups:
- Low Adherers: Subgroup of E-Moms Intervention group meeting less than and/or equal to 40% of expected number of days for logging weights and recording steps.
- Medium Adherers: Subgroup of E-Moms Intervention group meeting 40.1%-70% (3-5 days of engagement per week) of expected number of days for logging weights and recording steps.
- High Adherers: Subgroup of E-Moms Intervention group meeting greater than 70% (5 or more days of engagement per week) of expected number of days for logging weights and recording steps.
Arm/Group | Low Adherers | Medium Adherers | High Adherers | WIC Moms
Number analyzed (Participants) | 7 | 7 | 5 | 16
cm | 2.8 (1.4) | 0.96 (1.44) | -5.0 (1.7) | 0.62 (0.95)

3. Post Hoc Outcome: Changes in Waist Circumference of WIC Moms, WIC E-Moms Subgroups: High, Medium, and Low Adherers
Description: Changes in waist circumference from baseline (week 0) stratified by adherence to the E-Moms intervention and usual care (WIC Moms)
Time Frame: Baseline and 16 weeks
Population: All participants stratified by adherence to the E-Moms intervention and usual care (WIC Moms)
Measure: Mean (Standard Error); unit: cm
Arm/Group | Low Adherers | Medium Adherers | High Adherers | WIC Moms
Number analyzed (Participants) | 7 | 7 | 5 | 16
cm | 2.6 (2.2) | -2.5 (0.96) | -4.1 (2.6) | 0.99 (1.48)

4. Post Hoc Outcome: Changes in % Body Fat in WIC Moms, WIC E-Moms Subgroups: High, Medium, and Low Adherers.
Description: Changes in % body fat from baseline (week 0) stratified by adherence to the E-Moms intervention and usual care (WIC Moms).
Time Frame: Baseline and 16 weeks
Population: All participants stratified by adherence to the E-Moms intervention and usual care (WIC Moms)
Measure: Mean (Standard Error); unit: % body fat
Arm/Group | Low Adherers | Medium Adherers | High Adherers | WIC Moms
Number analyzed (Participants) | 7 | 7 | 5 | 16
% body fat | 1.1 (0.9) | 0.9 (0.9) | -2.5 (1.0) | 1.7 (0.6)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a year time span.
Description: Participant's were questioned by study staff at each study visit for any new or outstanding adverse event details.
Arm/Group | WIC E-Moms | WIC Moms
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/16
Other Adverse Events (participants affected / at risk) | 4/19 | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WIC E-Moms (N=19) | WIC Moms (N=16)
Cold (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Not Study Related
Viral infection (Infections and infestations) | 1 (1) | 1 (1) — Not Study Related
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Not Study Related
Flu (General disorders) | 1 (1) | 0 (0) — Not Study Related
Fatigue (General disorders) | 1 (1) | 0 (0) — Not Study Related

LIMITATIONS AND CAVEATS:
1) pilot and feasibility study (small sample size), 2) Variable adherence to the intervention, 3) greater lost to follow-up in the control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No